CLINICAL TRIAL: NCT00191607
Title: A Randomized Phase III Trial of Gemzar Versus Doxil With Crossover Treatment Option for Patients With Platinum-Resistant Ovarian, Fallopian Tube or Primary Peritoneal Cancer Undergoing Second or Third-Line Chemotherapy
Brief Title: A Randomized Trial for Patients With Platinum Resistant Ovarian, Fallopian or Primary Peritoneal Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6890; B9E-US-S301
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Genital Neoplasms, Female; Fallopian Tube Neoplasms; Ovarian Neoplasms; Pelvic Neoplasms; Peritoneal Neoplasms
MeSH Terms: conditions — Genital Neoplasms, Female; Fallopian Tube Neoplasms; Ovarian Neoplasms; Pelvic Neoplasms; Peritoneal Neoplasms | interventions — Gemcitabine; liposomal doxorubicin

INTERVENTIONS:
Drug: Gemcitabine
Drug: liposomal doxorubicin

SUMMARY:
This trial compares two chemotherapy agents for the treatment of recurrent ovarian, fallopian or primary peritoneal cancer in patients that have received and are no longer responding to Platinum based treatment. The purpose of this trial is to compare progression free survival between gemcitabine and liposomal doxorubicin. Progression free survival (PFS) is defined as the period from study entry until disease progression

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a documented pathologic diagnosis of epithelial ovarian (FIGO Stage I-IV), Fallopian tube or primary peritoneal carcinoma
* Patients must have received platinum-based, first-line chemotherapy but no more than one additional prior chemotherapy regimen. Patients must have recovered from the acute side effects of prior chemotherapy prior to enrollment in this trial.
* Patients must be considered to have platinum resistant disease based on the most recent platinum-based regimen given, i.e., have had a treatment-free interval in response to platinum of less than six months, or have progressed during platinum-based therapy
* Presence of measurable disease or CA-125 > or = to 100 on two separate occasions at least one week apart is required for this study
* Patient must have a Zubrod Performance Status of 0, 1 or 2

Exclusion

* Patients with a current diagnosis of epithelial ovarian tumor of low malignant potential (borderline carcinomas) are not eligible. Patients with a prior diagnosis of a low malignant potential tumor that was surgically resected and who have subsequently developed invasive adenocarcinoma are eligible.
* Patients who are currently undergoing abdominal or pelvic radiation therapy or patients who have received prior abdominal or pelvic radiation therapy are excluded.
* Patients with unstable angina or who have had a heart attack within the past six months are not eligible to participate.
* Patients who have received prior Gemzar or Doxil therapy are ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162
Dates: Start 2002-07; Study Completion 2005-11

PRIMARY OUTCOMES:
- Progression free survival (PFS) in patients who have failed one, but no more than two, prior treatments

SECONDARY OUTCOMES:
Secondary objectives:
Response rate
Duration of response
Time to treatment failure
Survival
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: CALL 1-877-CTLILLY (1-877-285-4559) OR 1-317-615-4559 MON-FRI 9AM-5PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri, United States

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274